CLINICAL TRIAL: NCT04827849
Title: The Effect of Nursing Care Based on Transition Theory of Meleis on Women's Adaptation to Motherhood and Perceptions of Newborn Baby
Brief Title: Theory of Meleis on Women's Adaptation to Motherhood and Perceptions of Newborn Baby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Duygu Yeşilfidan, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Duygu YEŞİLFİDAN, Filiz ADANA
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Newborn; Prenatal Care; Nursing Caries
Keywords: Nursing care; Prenatal; Newborn; Postpartum; Theory; Transition

STUDY DESIGN:
Intervention Model Description: Following recruitment, the pregnant women were divided into a study and a control group by randomization (1:2 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): The study group will be provided physical examination, pregnancy monitoring and training on transition to motherhood within the direction of nursing care based on Meleis's Transition Period Theory, in addition to the usual care provided by healthcare professionals.
  Interventions: Other: Structured education and follow-up
- Control group (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Other: Structured education and follow-up — The women in the intervention groups will administer a seven-session intervention program in addition to the routine care they will receive.
  The training including preparation practices for the transition with the mother, which is planned to last for 7 weeks encompassed providing the women with an educational programme that were created to increasing women's adaptation to motherhood and perceptions of newborn baby
  Nursing-recommended follow-up and physical examination of the pregnant woman will be performed at 28th and 34th week of pregnancy. In addition, postpartum and newborn follow-up, and mother-newborn physical examinations will be performed at the postpartum period.
  Arms: Experiment group

SUMMARY:
A randomised control trial will made to determine the effects of nursing care based on Meleis's Theory of Transition on Adaptation of Women to Motherhood and their Perception of New-born Infant

DETAILED DESCRIPTION:
Transition to motherhood, being one of the most important life incidents in the lives of women embodies the transition of role from a known situation to an unknown one. Being a special period in which women hold the role of motherhood together with the birth of the child; try to adapt the new role and reform relationship with the family members at the same time, transition to motherhood is a progressive period experienced by many women. Transition of woman to motherhood in a healthy manner will positively affect developing trust, achieving healthy communication with the infant, adapting to new lifestyle and fulfilling her responsibilities. Thus, transition to motherhood is quite significant both for mother and other family members and the new-born infant and needs to be discussed.

It is aimed in this research that effects of nursing care based on Meleis's Theory of Transition on Adaptation of Women to Motherhood and their Perception of New-born Infant shall be tested.

It will tested the hypotheses that there is no difference between the intervention and control groups of pregnant women after the intervention in terms of adaptation to pregnancy, adaptation to the postpartum period and newborn perception.

ELIGIBILITY:
Inclusion Criteria:

* Living in Aydın
* Between the ages of 18-35
* Have no children
* Gestational week is 28 weeks (beginning of 3rd trimester)
* Having a single pregnancy
* At least primary school graduate
* Not risky of pregnancy
* Have no chronic disease
* Can speak and write Turkish language

Exclusion Criteria:

* Having a history of mental and mental health problems
* With speech and hearing impairments
* Having a risky pregnancy
* Having multiple pregnancies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 79 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Adaptasion with pregnancy before intervention | 28th gestational weeks
  Adaptasion with pregnancy period will be evaluated with "Prenatal Self Evaluation Questionnaire".
  The scale was developed (1979) in order to evaluate the adaptation of women in the prenatal period to motherhood. The scale has 7 sub-dimensions. For the whole scale, a minimum of 79 and a maximum of 316 points can be obtained. Low scores show that adjustment to pregnancy is high.
Adaptasion with pregnancy after intervention | 34th gestational weeks
  The "Prenatal Self Evaluation Questionnaire" will be used to compare the fits to pregnancy between 28th and 34th weeks of gestation.
  The scale was developed (1979) in order to evaluate the adaptation of women in the prenatal period to motherhood. The scale has 7 sub-dimensions. For the whole scale, a minimum of 79 and a maximum of 316 points can be obtained. Low scores show that adjustment to pregnancy is high.
Mother-Neonatal Perception after birth | 3rd - 5th day after the birth
  Neonatal Perception Inventory (NPI-I) will be used to determine maternal- newborn perception.
  The scale was developed in 1971 to measure mothers' perception of their babies. It consists of two parts: the Neonatal Perception Inventory (NPI-I), applied in the first days after birth, and the NPI-II, administered one month after birth. In NPI-I and II of the scale, there are "Any Baby" and "Your Baby" forms, each containing six items (behaviors such as crying, feeding, sleeping, vomiting / drooling, pooping, eating and sleeping habits). It consists of 5-point Likert type 24 items.
Mother-Neonatal Perception after birth | 1st month after the birth
  Neonatal Perception Inventory (NPI-II) will be used to determine maternal- newborn perception.
  The scale was developed in 1971 to measure mothers' perception of their babies. It consists of two parts: the Neonatal Perception Inventory (NPI-I), applied in the first days after birth, and the NPI-II, administered one month after birth. In NPI-I and II of the scale, there are "Any Baby" and "Your Baby" forms, each containing six items (behaviors such as crying, feeding, sleeping, vomiting / drooling, pooping, eating and sleeping habits). It consists of 5-point Likert type 24 items.
Adaptasion to the postpartum period | 1st month after the birth
  The scale was developed (1981) to evaluate the adaptation of women in postpartum period to motherhood and is a 4-point Likert type with 82 items. There are 7 subscales that evaluate postpartum compliance of mothers. For the whole scale, a minimum of 82 and a maximum of 328 points can be obtained. Low scores indicate high postpartum adjustment.
Adaptasion to the postpartum period | 4th month after the birth
  The scale was developed (1981) to evaluate the adaptation of women in postpartum period to motherhood and is a 4-point Likert type with 82 items. There are 7 subscales that evaluate postpartum compliance of mothers. For the whole scale, a minimum of 82 and a maximum of 328 points can be obtained. Low scores indicate high postpartum adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Yeşilfidan, MsC, Study Chair — Aydın Adnan Menderes University, Faculty of Nursing, Devision Public Health Nursing
Locations (1):
- AydınAdnan Menderes University, Faculy of Nursing, Division Public Health Nursing, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.